CLINICAL TRIAL: NCT03964103
Title: Efficacy and Colon Attachment of gQ-lab Daily for Patients With Irritable Bowel Syndrome: Randomized, Double-blind, Placebo-controlled, Parallel-group Study
Brief Title: qQ-lab Daily-IBS for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: qQ-lab daily-IBS
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gQ-lab daily (Experimental)
  Interventions: Dietary Supplement: gQ-lab daily
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: gQ-lab daily — probiotics
  Arms: gQ-lab daily
Dietary Supplement: Placebo — powdered skim milk, lactose
  Arms: Placebo

SUMMARY:
* Primary purpose: To assess satisfaction with overall improvement in symptoms, including individual bowel symptoms, after 4 weeks of administration of gQ-lab to patients with irritable bowel syndrome (IBS).
* Secondary purposes: To assess the correlation between intestinal attachment and therapeutic effects of gQ-lab through the visual analog scale (VAS) assessment of each IBS-related symptom and measurement of changes in quality of life and fecal flora in the placebo group and gQ-lab group after 4 weeks of gQ-lab administration.

To assess safety, including adverse reactions, vital signs (including weight), physical examination, and changes in blood test results.

To examine the rate of positive gut quotient (gQ) values in patients diagnosed with IBS as per the ROME III criteria. Further, to examine how the ROME III-based symptom scale score compared with that of the quality of life scale in the gQ questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Korean men and women aged over 19 and 80
2. Patients with IBS meeting the ROME III criteria (Diagnosed with IBS with abdominal discomfort or abdominal pain in the past 3 months and meeting at least two of the following conditions: (1) improvement in defecation; (2) onset of symptoms associated with changes in stool frequency; (3) association with changes in stool form)
3. Patients who underwent colonoscopy in the past 5 years and have been confirmed to have no organ abnormalities
4. Women who are surgically infertile or fertile women who are negative during pregnancy diagnostic tests (urine or seron- hCG). Fertile women who have "almost no chance of becoming pregnant" during the study period owing to the use of appropriate contraception (e.g., oral contraceptive pills, IUD, double-barrier method, or hormone implants) or men who have agreed to this
5. People who have no problems in their nerves and mental systems and who can make their own doctors clear
6. The person who agreed in writing to this test

Exclusion Criteria:

1. Persons with hypersensitivity to probiotics
2. Pregnant or lactating women
3. People who have received other clinical trial drugs within the first 3 months of visit 1. (If the patient has received any other clinical trial drug within the past 3 months, contact the client's monitor to determine eligibility on a case-by-case basis.)
4. A person who believes that the participant is in a condition or situation in which participation in the clinical trial may be hazardous to the participant
5. Patients with severe congestive heart failure or severe angina
6. If the patient is diagnosed as having lactose intolerance or immunosuppression
7. Patients who are taking or taking medications (medicine for intestinal disorders, lactic acid bacteria) that may affect the test food, probiotics, or during the test period. However, if you are taking the drug, you can take the test after two weeks of abstinence.
8. If the systolic blood pressure measured at Visit 1 is greater than 160 mmHg or diastolic blood pressure is greater than 100 mmHg and hypertension is not controlled regardless of whether the medication is administered or not.
9. Patients with uncontrolled endocrine diseases (such as diabetes), metabolic diseases (e.g. secondary hyperlipidemia) or hypothyroidism (subjects with a history of hypothyroidism) should receive a stable thyroid hormone supplement for at least 4 weeks prior to visit 1 If you are on therapy, you can participate in this test only if the TSH level measured at Visit 2 is within the normal range.)
10. If kidney function is impaired at visit 1 (creatinine> 2.0 mg / dL) or nephrotic syndrome is observed
11. If the cancer has developed within the past 5 years (unless it is determined to be cured)
12. If there is a history of mental instability and drug / alcohol abuse within the past 5 years, or if major psychiatric illnesses are not adequately controlled and stabilized by medication
13. Visits 1 If you have taken mental nerve agents within the previous 3 months
14. If you take a systemic steroid preparation within 1 month before visit 1
15. Patients who underwent abdominal surgery except for appendectomy, hernia surgery, and cesarean section
16. Any person deemed inappropriate for the judgment of the clinician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Symptom questionnaire survey (VAS score) | 4 weeks
  To assess satisfaction with overall improvement in bowel symptoms, after 4 weeks of administration of GQ lab to patients with irritable bowel syndrome (IBS).
  The range of the VAS score is 1 to 10. The lower the value of the VAS score, the better. The value of the endpoint (4 weeks) is compared in the placebo group versus the treatment group.

IPD SHARING:
Plan to Share IPD: No